CLINICAL TRIAL: NCT03687437
Title: Diagnostic Accuracy of the Mean Platelet Volume in Oral Lichen Planus
Brief Title: Lichen Planus and Mean Platelet Volum
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Zakaria Ibrahium Mohammed, Lecturer of Oral Medicine and Periodontology, Cairo University, Egypt, Cairo University
Other Study IDs: Mai Zakaria
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Lichen Planus, Oral
Keywords: Oral lichen planus, mean platelet volume
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Complete blood count
  Other Names: Biopsy

SUMMARY:
70 patients with suspicious oral lichen planus; atrophic and bullous erosive forms will be included. The blood samples will be drawn between 08:00 and 09:00 AM, after a fasting period of 12 hours, and analysis were performed within 2 hours of the sampling. The MPV and other hematologic parameters will be measured in a blood sample. A surgical biopsy will be performed for histopathological assessment.

DETAILED DESCRIPTION:
70 patients with suspicious oral lichen planus; atrophic and bullous erosive forms will be included for conventional clinical examination under incandescent projected light. Using biopsy as a gold standard, all patients will be biopsied.

Blood Samples For all participants, the blood samples will be drawn between 08:00 and 09:00 AM, after a fasting period of 12 hours, and analysis were performed within 2 hours of the sampling. The MPV and other hematologic parameters will be measured in a blood sample that will be collected in tubes containing EDTA. Complete blood cell analysis will be performed in hematology laboratory, New Kasr Al-Aini Teaching Hospital, Faculty of Medicine, Cairo University. For reliable MPV measurement, the investigator will standardize the time delay between sampling and analysis to <2 hours for all patients.

Biopsy preparation A surgical biopsy will be performed for histopathological assessment. All clinically identified lesions underwent biopsies where specimens will be placed in 10% buffered formalin for fixation. Paraffin embedded material will be cut into 4 μm thick sections and will be stained with haematoxylin + eosin then submitted for histopathological evaluation by a senior oral pathologist blinded to the clinical findings.

Statistical analysis

The collected data will be entered through the SPSS version 18.0 software. Sensitivity, Specificity, Positive Predictive Value (PPV), Negative Predictive Value (NPV) and Accuracy were calculated for MPV. The results will be compared with histopathological results using Chi-Square test with p value set as < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria is suspected oral lichen planus, age 18-60

Exclusion Criteria:

* Foreseeable missing opportunity of follow-up examination, Pregnancy, heart-, pulmonary, liver- and kidney disease, chronic pain syndrome nursing, drug addiction, recent operations, and diseases like heart, metabolism, CNS, infectious, circulation, systemic, malignant and immune system affecting diseases as well as blood coagulation disorders and allergic reactions to pharmaceuticals and antibiotics

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients suspected to have oral lichen planus
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Complete blood count | Once at the time of the first visit
  blood sample between 08:00 and 09:00 AM and analysis to <2 hours for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Dalia El Rouby, PH, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Oral Medicine and Periodontology Department, Cairo
  - Faculty of Dentistry, Cairo University, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta S, Ghosh S, Gupta S. Interventions for the management of oral lichen planus: a review of the conventional and novel therapies. Oral Dis. 2017 Nov;23(8):1029-1042. doi: 10.1111/odi.12634. Epub 2017 Mar 3. PMID 28055124